CLINICAL TRIAL: NCT00787345
Title: General Surgery Residents Education in Maximum Barrier Precautions During Central Venous Catheter Placement: Effect of Simulation-Based Training
Brief Title: Simulation-based Training for Surgery Residents in Aseptic Techniques
Acronym: CVC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Hassan Khouli, MD, St. Luke's Roosevelt Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 08-094
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2008-05

CONDITIONS: Nosocomial Infections
Keywords: precaution technique during central venous catheter placement.
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery residents (Other): general surgery residents undergoing evaluation and training in MBP during CVC placement as per department policy are eligible for the study.
  Interventions: Other: simulation based training

INTERVENTIONS:
Other: simulation based training — simulation based training in aseptic techniques that included specified AT categories

SUMMARY:
Central line associated bloodstream infection (CL-ABI) is an important and preventable cause of nosocomial infections and is responsible for considerable morbidity and mortality The Centers for Disease Control have published guidelines for the prevention of CL-ABI that represent a collaborative effort by a multidisciplinary coalition of professional organizations that provide evidence based recommendations to prevent catheter related infections [5]. The interventions emphasize five distinct practices, including: education and training of healthcare providers who place and care for catheters, utilizing maximum sterile barrier precautions during catheter placement.

DETAILED DESCRIPTION:
Central line associated bloodstream infection (CL-ABI) is an important and preventable cause of nosocomial infections and is responsible for considerable morbidity and mortality. It is estimated that 5 to 26% of patients experience an infectious complication from their central venous catheter [1]. In the United States, it is estimated that nearly 50,000 patients develop central line associated bloodstream infections in the ICUs annually, at a rate of approximately 5 infections per 1000 catheter days [2] and as many as 15,000 deaths annually. Central line associated bloodstream infections are also associated with increased hospital and ICU lengths of stay in the ICU (2). Estimates of the cost of CL-ABI to hospitals range from $25,000 to $65,000 per patient [3, 4].

The Centers for Disease Control have published guidelines for the prevention of CL-ABI that represent a collaborative effort by a multidisciplinary coalition of professional organizations that provide evidence based recommendations to prevent catheter related infections [5]. The interventions emphasize five distinct practices, including: education and training of healthcare providers who place and care for catheters, utilizing maximum sterile barrier precautions during catheter placement, skin preparation using 2% chlorhexidine, avoiding routine replacement of central lines as a strategy to reduce infection, and using antiseptic or antibiotic coated lines in the event that infection rates remain high despite adherence to the above measures [5].

Several studies have demonstrated impressive reductions in CL-ABI from the application of these strategies, ranging from 18 to 100% reductions and realizing significant reductions in mortality and cost [2]. The simple introduction of maximum sterile barrier precautions to insert central lines has been observed to dramatically reduce infection rates for over a decade [6]. However, the CDC's guidelines, despite their seeming simplicity, have been found to be frequently insufficiently applied, whether by ignorance or omission [2].

In the past 12 months there have been a total 24 documented central venous line (CVL) infections at SLRHC with cumulative rate of infection of 3.8 per 1000 central line days. These infection rate figures are above the benchmark experience. For SLRHC the cost incurred over the past 12 months is estimated to be $1,080,000.

Training and education of healthcare personnel and the utilization of maximum sterile precautions are two important areas. Residents still most frequently learn central line placement techniques by the "see one, do one, teach one" method, which by its very definition allows for a multitude of techniques in practice. While this teaching theoretically includes the utilization of maximal sterile precautions for central line placement, the focus of teaching, and of residents' anxieties, is most often focused on the proper placement of the line, not the sterile technique used to place it. Guzzo et al found that mentors of trainees performing CVC placements in both emergent and non-emergent situations were significantly less likely to consistently utilize maximum sterile precautions [8]. Furthermore, in a study of a video-based training on sterile technique in CVC insertion in a trauma resuscitation unit that evaluated only non-emergent CVC placements, a total of 5 cases of central- catheter- related bacteremia were reported on just 68 patients, and even with video based training, 26% of residents continued to have infractions in their compliance with sterile precautions [9].

Medical simulators allow residents to practice skills in a realistic and interactive environment that minimizes risk to patients. Studies have found simulation to be an effective means for teaching skills as diverse as ACLS and airway management to laparoscopic surgical skills [10,11,12]. Additionally, the use of audio-visual equipment in a medical simulator to record a resident's performance gives valuable firsthand feedback that is otherwise not available, as it allows residents to visualize their own missteps [13]. This is hypothesized to be of particular value in the proper acquisition of physical skills such as maximum sterile precautions.

With this in mind, the Department of Surgery has recently approved a training policy in aseptic technique during central venous access placement (see attached copy). All GS residents will be trained in MBP techniques in the Sim Lab. Training will include baseline assessment of residents skills in maintaining maximum sterile precautions using a standardized scoring tool, videotape training, short exam, and individual simulated debriefing on performance of correct MBP with follow up assessment and training as needed.

We plan to collect data prospectively on all GS residents who will undergo evaluation and training in maximum barrier precaution during CVC placement. Data will be reviewed and analyzed for future research publication

C METHODS:

I. Inclusion criteria:

General Surgery (GS) residents will be undergoing evaluation and training in MBP according to their department training policy.

II. Design:

A. All GS residents undergoing evaluation and training in MBP during CVC placement as per department policy are eligible for the study.

B. All data collected for the purpose of Education and Quality Improvement on all GS residents, who are undergoing evaluation and training (as per standard department policy) in MBP during CVC placement will be reviewed and analyzed after being deidentified for the purpose of this study.

C. Waiver of Subject informed consent and HIPPA authorization is requested as this is a minimal risk study and the data and thus conclusions would be greatly improved by using the data from all subjects. There could be a selection bias if we only used the data from the residents who felt they had done a good job. Other criteria needed to waiver of subject informed consent and HIPPA authorization are listed below:

1. Minimal risk study: This is an observational, non-interventional study. The research part of the study is the prospective data collection for the purpose of analysis of the aggregate data and possible publication. Training of residents in MBP as per described protocol is set according to approved hospital policy for the purpose of quality improvement. The only risk to the subject is the potential loss of confidentiality, and the investigators will minimize that risk by deidentifying the data as described below in section III (Confidentiality) and all research data will be deleted once the six month follow-up has been completed
2. There is no reason to believe that waiving the informed consent will affect the rights and welfare of the subjects enrolled since these subjects will not be identified by name or any form of identity. Also, all subjects will be informed that final project results that include all subjects will be reviewed as a group and no personal identifications will be included in the results.
3. This research may not be carried out without the waiver as the results and thus conclusions would be greatly improved by using the data from all subjects. There could be a selection bias if we only used the results from the residents who felt they had done a good job
4. This research may benefit the subjects directly by understanding the limitations of previous training (or lack of) in MBP if any noted after analyzing the results, and is likely to yield generalizable knowledge that would be of benefit for subjects with similar conditions.
5. This area of research is directly related to the condition of any potential subjects who might not be able to give consent
6. Whenever appropriate the subjects will be provided with additional pertinent information after participation as it has been stated in the protocol
7. Protections will be taken to protect the confidentiality of subjects as outlined below in the Confidentiality section D. Information sheet will be provided to all residents participating in this project explaining the purpose of this project, confidentiality protection when data is potentially reported, and E. GS residents may have repeated performance (3-6 months) in MBP technique for central line placement individually at the discretion of their residency program director. If so, data collected will be analyzed and reviewed.

III. Confidentiality:

All aggregate data will be kept secured as part of the research database and will be password protected. No supervisor will have access to this aggregate data and he / she will not be able to compare any individual resident's performance to the rest of the group in the database.

All sessions in the sim lab are videotaped automatically. All videotapes sessions titles are not identified by name but coded (i.e sim session medical code session 6 June 08). All videotapes are reviewed periodically and deleted except for few that are kept for educational purpose. These videotapes are identified by subject study number and phase only (i.e. CVLN 01 phase 1). In this project, videotaping of all subjects performances is for the purpose of training, and quality improvement. The research part of this project involves review of the data collected by the instructor on the assessment tool and is unrelated to videotaping.

IV. Data Analysis The overall performance score of MBP technique, including the overall maximum and the seven components will be analyzed. The effects of simulation based training on performance, realized in performance score improvement over baseline, will be evaluated using Wilcoxon signed-rank test. A p-value less than 0.05 will be considered as statistically significant

ELIGIBILITY:
Inclusion Criteria:

* General surgery residents will be undergoing evaluation and training in MBP according to their department training policy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Primary outcome: General surgery residents performance in maximal barrier precaution (MBP) technique during central venous catheter (CVC) placement | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Khouli, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (2):
- United States (2):
  - SLRH, New York, New York
  - St.Luke's Roosevelt Hospital, New York, New York

REFERENCES:
- [Background] McGee DC, Gould MK. Preventing complications of central venous catheterization. N Engl J Med. 2003 Mar 20;348(12):1123-33. doi: 10.1056/NEJMra011883. No abstract available. PMID 12646670
- [Background] Eggimann P. Prevention of intravascular catheter infection. Curr Opin Infect Dis. 2007 Aug;20(4):360-9. doi: 10.1097/QCO.0b013e32818be72e. PMID 17609594
- [Background] Posa PJ, Harrison D, Vollman KM. Elimination of central line-associated bloodstream infections: application of the evidence. AACN Adv Crit Care. 2006 Oct-Dec;17(4):446-54; quiz 456. doi: 10.4037/15597768-2006-4009. PMID 17091045
- [Background] Bull DA, Neumayer LA, Hunter GC, Sethi GK, McIntyre KE, Bernhard VM, Putnam CW. Improved sterile technique diminishes the incidence of positive line cultures in cardiovascular patients. J Surg Res. 1992 Feb;52(2):106-10. doi: 10.1016/0022-4804(92)90287-a. PMID 1740929
- [Background] Pronovost P, Needham D, Berenholtz S, Sinopoli D, Chu H, Cosgrove S, Sexton B, Hyzy R, Welsh R, Roth G, Bander J, Kepros J, Goeschel C. An intervention to decrease catheter-related bloodstream infections in the ICU. N Engl J Med. 2006 Dec 28;355(26):2725-32. doi: 10.1056/NEJMoa061115. PMID 17192537
- [Background] Guzzo JL, Seagull FJ, Bochicchio GV, Sisley A, Mackenzie CF, Dutton RP, Scalea T, Xiao Y. Mentors decrease compliance with best sterile practices during central venous catheter placement in the trauma resuscitation unit. Surg Infect (Larchmt). 2006 Feb;7(1):15-20. doi: 10.1089/sur.2006.7.15. PMID 16509781
- [Background] Xiao Y, Seagull FJ, Bochicchio GV, Guzzo JL, Dutton RP, Sisley A, Joshi M, Standiford HC, Hebden JN, Mackenzie CF, Scalea TM. Video-based training increases sterile-technique compliance during central venous catheter insertion. Crit Care Med. 2007 May;35(5):1302-6. doi: 10.1097/01.CCM.0000263457.81998.27. PMID 17414726
- [Background] Wayne DB, Siddall VJ, Butter J, Fudala MJ, Wade LD, Feinglass J, McGaghie WC. A longitudinal study of internal medicine residents' retention of advanced cardiac life support skills. Acad Med. 2006 Oct;81(10 Suppl):S9-S12. doi: 10.1097/00001888-200610001-00004. PMID 17001145
- [Background] Mayo PH, Hackney JE, Mueck JT, Ribaudo V, Schneider RF. Achieving house staff competence in emergency airway management: results of a teaching program using a computerized patient simulator. Crit Care Med. 2004 Dec;32(12):2422-7. doi: 10.1097/01.ccm.0000147768.42813.a2. PMID 15599146
- [Background] Murray D. Clinical simulation: measuring the efficacy of training. Curr Opin Anaesthesiol. 2005 Dec;18(6):645-8. doi: 10.1097/01.aco.0000188419.77140.1a. PMID 16534306
- [Background] Savoldelli GL, Naik VN, Park J, Joo HS, Chow R, Hamstra SJ. Value of debriefing during simulated crisis management: oral versus video-assisted oral feedback. Anesthesiology. 2006 Aug;105(2):279-85. doi: 10.1097/00000542-200608000-00010. PMID 16871061
- [Background] Shannon RP, Patel B, Cummins D, Shannon AH, Ganguli G, Lu Y. Economics of central line--associated bloodstream infections. Am J Med Qual. 2006 Nov-Dec;21(6 Suppl):7S-16S. doi: 10.1177/1062860606294631. PMID 17077414